CLINICAL TRIAL: NCT03129750
Title: Safety and Efficacy of the Drug Coated Balloon (DCB) for the Treatment of the Superficial Femoral Artery (SFA) Ischemic Vascular Disease in Symptomatic Patients Presenting With TASC C and D Lesions: a Pilot Study
Brief Title: Safety and Efficacy of DCB for the Treatment of SFA Ischemic Vascular Disease in Patients With TASC C and D Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO26
Record Dates: First submitted 2016-09-30; First posted 2017-04-26 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: PAD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Drug Coated Balloon — Peripheral PTA with a drug coated balloon

SUMMARY:
The study is aimed at collecting preliminary safety and efficacy data related to the use of Drug Coated Balloon (DCB) technology for the treatment of symptomatic Superficial Femoral Artery (SFA) ischemic vascular disease in patients presenting with long lesions.

The present clinical evaluation is intended as a prospective observational data collection of patient treatment in full accordance with institution standard practice and utilizing an approved (CE marked) DCB currently available on the market.

DETAILED DESCRIPTION:
The present study is designed as a prospective, open label, observational study.

The study will collect information about the medical care patients receive during their planned procedure. No additional testing or procedures will be done.

Patients elected for endovascular revascularization with DCB will be asked their written consent to the use of their personal data.

Revascularization will be performed as per standard procedure of the sites. After discharge all patients will attend clinic visits at 30 days (±14 days), 6 months (±30 days), 12 months (±30 days), 24 and 36 months (±30 days). Angiographic follow-up will be performed in symptomatic patients, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Documented obstructive ischemic, symptomatic arterial disease in the femoral-popliteal arteries according to Rutherford Category 2, 3 or 4
2. Target lesion consists of a single solitary or multiple adjacent de novo or re-stenotic lesions (non-in-stent) with diameter stenosis ≥ 70% by visual estimate and cumulative lesion length ≥ 15 cm
3. Target vessel is the superficial femoral artery and/or popliteal artery (P1-2-3)
4. Life expectancy >1 year in the Investigator's opinion
5. Written informed consent

Exclusion Criteria:

1. Patient unwilling or unlikely to comply with FU schedule
2. Administration of local or systemic thrombolytic therapy within 48 hours prior to the index procedure
3. Known allergies or sensitivities to heparin, aspirin, other anticoagulant/antiplatelet therapies, and/or paclitaxel
4. Additional planned cardiac or peripheral percutaneous or surgical intervention including CABG within 30 days following the study procedure
5. ≥15 cm long inflow lesion (≥50% DS)
6. Failure to successfully treat < 15 cm long inflow lesion in the ipsilateral Iliac artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients with ischemic vascular disease presenting with TASC C and D.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Rate of primary patency | 12 months after percutaneous treatment
  Primary patency is defined as freedom from the combined endpoints of clinically-driven target lesion revascularization (TLR) and >50% restenosis in the treated lesion.

SECONDARY OUTCOMES:
composite of all Major Adverse Events (MAE) | 24 months after percutaneous treatment
  Incidence of the composite of all Major Adverse Events (MAE) through 24 months
Incidence of Major Adverse Events (MAE) | 36 months after percutaneous treatment
  Incidence of Major Adverse Events (MAE) through 36 months
Clinical improvement as assessed by Rutherford Class changes | 6, 12, 24 and 36 months vs baseline
  Clinical improvement as assessed by Rutherford Class changes

OTHER OUTCOMES:
Rate of instrumental restenosis | Post-Procedure
  Rate of instrumental restenosis as determined by duplex ultrasound Peak Systolic Velocity Ratio (PSVR) > 2 post-index procedure evaluated by an independent core lab
Procedural success rate | end of percutaneous procedure
  Rate of procedural success in the absence of peri-procedural complications
Walking capacity and quality of life | 6, 12, 24 and 36 months post-procedure
  walking capacity as assessed by walking impairment questionnaire (WIQ), and 6 minutes' walk test
Rate of instrumental restenosis | 12, 24 and 36 months
  Rate of instrumental restenosis as determined by duplex ultrasound Peak Systolic Velocity Ratio (PSVR) > 2 evaluated by an independent core lab
Quality of Life | 6, 12, 24 and 36 months post-procedure
  quality of life assessed by EQ5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Micari, MD, Principal Investigator — Maria Cecilia Hospital
Locations (10):
- Italy (10):
  - Casa di Cura Montevergine, Mercogliano, Avellino
  - ICLAS, Rapallo, Genova
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Santa Maria Hospital, Bari
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Città di Lecce Hospital, Lecce
  - Policlinico Federico II, Napoli
  - Maria Eleonora Hospital, Palermo
  - Azienda Policlinico Umberto I di Roma, Roma
  - Maria Pia Hospital, Torino

IPD SHARING:
Plan to Share IPD: No